CLINICAL TRIAL: NCT06729437
Title: Effectiveness of Transcranial Direct Current Stimulation on Functionality and Pain in Individuals with Patellar Tendinopathy: Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation on Functionality and Pain in Individuals with Patellar Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-FIS-3100133
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Patellar Tendinopathy
Keywords: patellar tendinopathy; transcranial direct current stimulation; therapeutic exercise; eccentric exercise
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants will undergo an 8-week intervention of supervised eccentric exercise by a physiotherapist (3 sessions/week). During the first 4 weeks, real tDCS will be administered at a rate of 3 sessions per week (12 in total) as an adjunct to exercise . A direct current of 1.5 mA will be applied for 20 minutes to the primary motor cortex (M1) during each session of eccentric exercises. Additionally, all participants will perform the eccentric exercise program on the remaining weekdays at home unsupervised.
  Interventions: Other: tDCS + Therapeutic eccentric exercise
- Sham group (Placebo Comparator): Participants will undergo an 8-week intervention of supervised eccentric exercise by a physiotherapist (3 sessions/week). During the first 4 weeks, sham tDCS will be administered at a rate of 3 sessions per week (12 in total) as an adjunct to exercise. The current will be interrupted after 30 seconds. Additionally, all participants will perform the eccentric exercise program on the remaining weekdays at home unsupervised.
  Interventions: Other: Sham tDCS + Therapeutic eccentric exercise

INTERVENTIONS:
Other: tDCS + Therapeutic eccentric exercise — A direct current of 1.5 mA will be applied for 20 minutes to the primary motor cortex (M1) during each session of eccentric exercises.
  Arms: Experimental group
Other: Sham tDCS + Therapeutic eccentric exercise — The current will be interrupted after 30 seconds.
  Arms: Sham group

SUMMARY:
The aim of the present study is to investigate the effectiveness of transcranial direct current stimulation (tDCS) prior to a therapeutic eccentric exercise program on parameters related to pain and functionality in individuals with patellar tendinopathy. For this purpose, participants will be randomly divided into two groups: i) experimental group, receiving tDCS prior to a therapeutic exercise program; and ii) control group, receiving sham tDCS and a therapeutic exercise program. The interventions will last for 8 weeks. Additionally, four assessments will be conducted (baseline, week 4, week 8 and week 12). The variables studied are related to pain, functionality, muscle activity and strength, proprioception, and quality of life.

DETAILED DESCRIPTION:
Patellar tendinopathy is a painful condition affecting the anterior portion of the knee, commonly exacerbated by activities putting pressure on the patellofemoral joint. It remains a challenge for the healthcare system, not only due to its high prevalence, but also because of its high persistence and negative consequences. Although therapeutic exercise has been widely studied as a treatment strategy, eccentric exercise protocols, while effective, often require long application periods, which may affect treatment adherence. Additionally, eccentric exercise is pain-provoking and its therapeutic benefits for pain relief and functional improvement are controversial when used during the competitive season. More adaptable and personalized treatment strategies could enhance clinical outcomes and treatment adherence in patients with patellar tendinopathy. In this context, interventions combining exercise with other techniques have been proposed. However, existing evidence does not definitively determine the optimal approach for combining conservative treatment options to maximize benefits.

An emerging therapeutic approach combines Transcranial Direct Current Stimulation (tDCS) with therapeutic exercise protocols. tDCS involves the application of weak direct current to specific cortical areas, aiming to modulate brain excitability. This non-invasive method offers painless, selective, and focal stimulation with minimal side effects. Research increasingly supports the effectiveness of integrating tDCS with exercise for patellar tendinopathy, offering the potential to amplify exercise effects by modulating brain excitability. However, to date, no study has investigated the impact of tDCS combined with eccentric exercise on variables related to function and pain in patellar tendinopathy individuals.

Therefore, the aim of this study is to investigate the effectiveness of tDCS prior to a therapeutic eccentric exercise program on parameters related to pain and functionality in individuals with patellar tendinopathy.

This study is a randomized clinical trial in which two groups will participate, with different interventions: i) Experimental group: tDCS + Therapeutic eccentric exercise; and ii) Control group: Sham tDCS + Therapeutic eccentric exercise. The interventions will last for 8 weeks. Participants will be evaluated in four moments, at baseline, week 4, week 8 and week 12. The variables studied are related to pain, functionality, muscle strength and activity, proprioception, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Diagnosis of patellar tendinopathy (VISA-P score of 80 or lower).
* Pain lasting more than 3 months.

Exclusion Criteria:

* Previous knee surgery.
* Corticosteroid injection in the previous 6 weeks.
* Systemic inflammatory, autoimmune, or rheumatic diseases.
* Cognitive or behavioural issues that hinder comprehension and adherence to the intervention.
* Any neurological disease.
* Neoplastic disease.
* Subjects presenting contraindications for tDCS (Thair et al., 2017), including: personal and family history of epilepsy, metallic implants in the head, implanted medication pump, pacemaker, recurrent headaches, skin conditions (psoriasis, eczema), or major head surgeries, pregnancy, heart diseases, and various medications (psychotropic or antihistamines).
* Subjects must not have undergone pharmacological treatment or knee physical rehabilitation programs for a period of 1 year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Knee functionality | 5 minutes
  The Victorian Institute of Sport Assessment-Patella (VISA-P) is a questionnaire to assess the severity of patellar tendinopathies. It consists of 8 items with a rating range from 0 to 100. The optimal state would correspond to a score of 100.

SECONDARY OUTCOMES:
Pain intensity | 2 minutes
  The single-leg squat pain provocation test is used to monitor the response to previous loading in athletes with patella tendinopathy. A visual analogue scale (VAS) will be used to determine pain intensity during the test. A score of 0 points indicates no pain and 10 points is the worst imaginable pain.
Health-related quality of life | 2 minutes
  The EuroQol 5 dimensions (EQ-5D) test is an instrument which evaluates the generic quality of life. Scores range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Muscle strength | 10 minutes
  Maximum voluntary isometric contraction of the quadriceps, hamstrings, and hip abductors will be measured using a force sensor connected to the corresponding software (Chronojump Boscosystem). Higher values indicate greater muscle strength.
Electromyographic activity of lower limb muscles | 5 minutes
  Electromyographic activity during maximum voluntary isometric contraction of the rectus femoris, vastus lateralis, vastus medialis, biceps femoris, and semitendinosus muscles, using electromyography, will be registered.
Muscle flexibility | 5 minutes
  Knee joint range of motion will be measured in flexion and extension using a goniometer. Higher values indicate greater muscle flexibility.
Muscle tone | 5 minutes
  The biomechanical and viscoelastic properties of the muscle tissue will be evaluated using a non-invasive myometer, MyotonPRO (Myoton AS, Tallinn, Estonia). The patellar tendon, rectus femoris, vastus medialis, vastus lateralis, semitendinosus, and biceps femoris will be assessed. Higher values may indicate greater muscle stiffness or tone.
Proprioception | 5 minutes
  Proprioception will be assessed using the active knee repositioning test with an inclinometer. The difference between the target angle and the obtained angle will be registered. A smaller difference between the angles indicates better knee proprioception.
Patient global perception of change | 1 minute
  The Patient Global Impression of Change Scale (PGIC) will be filled out. It consists of 7 points, with options ranging from "1=much better" to "7=much worse".

CONTACTS AND LOCATIONS:
Overall Officials: Marta Inglés, Dr, Principal Investigator — Univeristy of Valencia
Locations (1):
- Faculty of Physiotherapy, University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang Y, Jetton TL, Zimmerman EC, Najafi H, Berner DK, Matschinsky FM, Magnuson MA. Effects of glucose on insulin secretion, glucokinase activity, and transgene expression in transgenic mouse islets containing an upstream glucokinase promoter-human growth hormone fusion gene. Diabetes. 1994 Sep;43(9):1138-45. doi: 10.2337/diab.43.9.1138. PMID 8070614
- [Background] Cosca DD, Navazio F. Common problems in endurance athletes. Am Fam Physician. 2007 Jul 15;76(2):237-44. PMID 17695568
- [Background] Vairel EG. [Enzyme systems and the means to study them]. Biol Med (1971). 1973 Dec;2(2):123-39. No abstract available. French. PMID 4620252
- [Background] Hernandez-Sanchez S, Hidalgo MD, Gomez A. Cross-cultural adaptation of VISA-P score for patellar tendinopathy in Spanish population. J Orthop Sports Phys Ther. 2011 Aug;41(8):581-91. doi: 10.2519/jospt.2011.3613. Epub 2011 Jul 12. PMID 21765223
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845
- [Background] Peers KH, Lysens RJ. Patellar tendinopathy in athletes: current diagnostic and therapeutic recommendations. Sports Med. 2005;35(1):71-87. doi: 10.2165/00007256-200535010-00006. PMID 15651914
- [Background] McKittrick JE, Henrikson J, Iwasiuk GW. Indications for contralateral carotid endarterectomy: role of the noninvasive laboratory. Am J Surg. 1980 Aug;140(2):206-8. doi: 10.1016/0002-9610(80)90006-9. PMID 7406123
- [Background] Dugois P, Amblard P, Gagnaire J, Imbert R. [Leg abscesses in stages after phlebosclerosus: complication of a septicemia of dental origin]. Bull Soc Fr Dermatol Syphiligr. 1968;75(4):518-20. No abstract available. French. PMID 5702643
- [Background] Vander Doelen T, Jelley W. Non-surgical treatment of patellar tendinopathy: A systematic review of randomized controlled trials. J Sci Med Sport. 2020 Feb;23(2):118-124. doi: 10.1016/j.jsams.2019.09.008. Epub 2019 Sep 13. PMID 31606317
- [Background] Visnes H, Hoksrud A, Cook J, Bahr R. No effect of eccentric training on jumper's knee in volleyball players during the competitive season: a randomized clinical trial. Clin J Sport Med. 2005 Jul;15(4):227-34. doi: 10.1097/01.jsm.0000168073.82121.20. PMID 16003036
- [Background] Srivastava RA, Schonfeld G. Use of riboprobes for northern blotting analysis. Biotechniques. 1991 Nov;11(5):584, 586, 588. PMID 1725109